CLINICAL TRIAL: NCT01532505
Title: A Randomized Study Comparing Low Dose Vasopressin Infusion or Placebo on Near Infrared Spectroscopy Tissue Oxygen Saturation and the Vascular Occlusion Test in Cardiac Surgery Patients During Cardiopulmonary Bypass: A Pilot Study
Brief Title: Effect of Vasopressin on Tissue Oxygen Saturation in Cardiac Surgery Patients During Cardiopulmonary Bypass
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mohamed Ismail (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, Mohamed Ismail, Principal investigator, London Health Sciences Centre
Organization: London Health Sciences Centre (Other)
Other Study IDs: 18511
Record Dates: First submitted 2012-01-19; First posted 2012-02-14 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Hypotension; Poor Peripheral Perfusion
Keywords: cardiopulmonary bypass; Postcardiotomy vasodilatory shock; Microcirculation; Catecholamines; Vasopressin
MeSH Terms: conditions — Hypotension; Diabetes Insipidus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this research is to compare the effect of a low dose Vasopressin infusion or placebo during cardiopulmonary bypass on vasopressor requirements, hemodynamics and tissue oxygen saturation and its recovery using tNIRS and vascular occlusion test (VOT) in elective on pump cardiac surgery patients using a non-invasive near infrared spectrometry (NIRS) machine. The clinical implications are that NIRS may permit earlier, non-invasive detection of significant physiologic derangements and allow more accurate and timely titration of medications, fluids and surgical intervention. The use of a low dose vasopressin seems to be preventive for the incidence of observed post-cardiotomy vasodilatory shock and may improve the function of microcirculation that will be assessed using VOT and tNIRS. Finally, it may decrease both catecholamine dose and duration of their administration, it is considered as a useful agent for decreasing all heir side-effects

DETAILED DESCRIPTION:
In our double blind randomized study 40 patients undergoing cardiac surgery will be randomly divided in two groups. The group A who will be infused with 2 IU/hr. vasopressin and the group B who will be infused with normal saline (placebo) intraoperatively starting at the time we give I.V. Heparin, throughout CPB and infusion will be ended when we give the Protamine after coming off bypass. VOTs will be measured at the following time points: Pre-induction of anesthesia, post-induction of anesthesia and at 30 minute intervals during the cardiopulmonary bypass. And we will select cases that are expected to have a longer CPB time such as Redo CABG, CABG + valve replacement, double valve replacement, Bentall procedure and Mitral valve repair with mini thoracotomy.

Measurements of mean artery pressure (MAP), central venous pressure (CVP), ejection fracture (EF), heart rate (HR), mean pulmonary artery pressure (MPAP), cardiac index (CI) will be performed before, during, and after the operation. The requirements of catecholamine support (eg. phenylephrine, epinephrine, vasopressin, norepinephrine, and dopamine) during CPB and for first 24 hours postoperatively, urine-output, blood-loss, and the requirements in blood, plasma and platelets for the first 24 hours will be included in the data collected.

The purpose of the present study is to quantify the micro-oxygenation parameters in patients undergoing cardiac surgery with CPB, to investigate the relationship of micro-oxygenation and macro-perfusion parameters, to investigate the relationship of NIRS parameters and to evaluate the association between micro-oxygenation parameters and outcome using VOT and comparing the degree of falling of re-perfusion slope.

We hypothesize that the administration of a low dose vasopressin will reduce both the incidence and severity of vasoplegia and it will maintain the normal vasomotor reactivity during cardiopulmonary bypass and this will reduce the total requirements of alpha-adrenergic agonists specially Phenylephrine. That will reduce the risks of the use of high dose of Phenylephrine and other inotropes, such as gut ischemia and end organ damage.

Vascular Occlusion Test (VOT)

* After the tissue oximetry probe is applied to the skin the oximeter machine records a baseline value.
* A pneumatic cuff (blood pressure cuff) is placed over the brachial artery of the same arm above the elbow and inflated to 50 mmHg above systolic blood pressure. The cuff remains inflated for 5 minutes. The oximeter machine is continuously recording StO2 values and other pertinent technical information such as quality of the signal and events marked by the user.
* After 5 minutes the cuff is quickly deflated and StO2 measurements continue to be recorded until back to baseline.
* VOTs will be measured at the following time points:
* Pre-induction of anesthesia
* Post-induction of anesthesia
* At 30 minute intervals during the cardiopulmonary bypass

Several measurements and calculations will be made from the recorded data:

* Baseline tissue oxygen saturation (StO2baseline) at time (t) = 0
* Lowest StO2 reached after vascular occlusion (StO2nadir) and at what time
* Occlusion slope: defined as = (StO2baseline - StO2nadir/tbaseline - tnadir)
* After cuff release, time at which baseline StO2 was reached (StO2recovery)
* Reperfusion slope: defined as = (StO2recovery - StO2nadir/trecovery - tnadir)
* ∆StO2: defined as = (StO2peak - StO2baseline)
* Peak StO2 reached after cuff release and at what time

Measurements of mean artery pressure (MAP), central venous pressure (CVP), ejection fracture (EF), heart rate (HR), mean pulmonary artery pressure (MPAP), cardiac index (CI) will be performed before, during, and after the operation. The requirements of catecholamine support (eg. phenylephrine, epinephrine, vasopressin, norepinephrine, dopamine) during CPB and for first 24 hours postoperatively, urine-output, blood-loss, and the requirements in blood, plasma and platelets for the first 24 hours will be included in the data collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult, elective cardiac surgery patients with the use of cardiopulmonary bypass (CPB)

Exclusion Criteria:

* Age less than 18 years
* Contraindication to pneumatic cuff inflation (arteriovenous fistula, previous mastectomy, injury to arm)
* Pregnancy
* Significant peripheral vascular disease of the arms*
* Emergency surgery
* Uncured cancer during chemotherapy
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable patients coming from home for elective cardiac surgery are eligible to participate
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
VOT assessment of microcirculation | day one
  change in reperfusion slope of VOT will be assessed each 30 min during CPB and compared between vasopressin and placebo patients

CONTACTS AND LOCATIONS:
Overall Officials: MOHAMED ISMAIL, MD,MSc, Principal Investigator — London HSC; JOHN MURKIN, MD, FRCPC, Study Director — London HSC
Locations (1):
- University Hospital, LHSC, London, Ontario, Canada

REFERENCES:
- [Background] Peripheral Tissue Oxygen Saturation (SaO2) Monitoring and the Vascular Occlusion Test in Cardiac Surgery: A Pilot Study. Smith R, Murkin J, Granton J, Guo LR, McKenzie FN, Min F, Zhang R. ASA Chicago, Oct 15-19, 2011, Anesthesiology 2011 A278.
- [Background] Papadopoulos G, Sintou E, Siminelakis S, Koletsis E, Baikoussis NG, Apostolakis E. Perioperative infusion of low- dose of vasopressin for prevention and management of vasodilatory vasoplegic syndrome in patients undergoing coronary artery bypass grafting-A double-blind randomized study. J Cardiothorac Surg. 2010 Mar 28;5:17. doi: 10.1186/1749-8090-5-17. PMID 20346182